CLINICAL TRIAL: NCT00712387
Title: A National, Prospective,Randomised, Single Blinded Controlled Trial of Proficiency- Based Simulation Training for General Surgical Trainees
Brief Title: Trial of Proficiency- Based Simulation Training for General Surgical Trainees
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: Health Service Executive (Unknown)
Responsible Party: Professor Anthony G Gallagher, National Surgical Training Centre, Royal College of Surgeons, Ireland
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: RCSI2
Record Dates: First submitted 2008-07-07; First posted 2008-07-10 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Education; Training; Computer Simulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (No Intervention): General surgical trainees who will receive the 'traditional' training programme; i.e. will receive whatever clinical training on a patient their supervising consultant deems appropriate. This is the way junior surgeons are currently trained. They will also receive the standard didactic teaching on the School for Surgeons e-learning resource.
- B (Active Comparator): Surgical trainees who are assigned to the 'proficiency-based progression' training programme. These trainees will be required to train on the virtual reality simulator (Lap Sim™) for a laparoscopic cholecystectomy. Trainees will have objectively set goals to reach on the simulator and will have to demonstrate proficiency before they are permitted to progress to the next, more challenging level. Group B will also receive the standard School for Surgeons instruction but, unlike Group A, they will have to demonstrate proficiency on the didactic module before they progress to the operating theatre
  Interventions: Behavioral: LapSim simulator

INTERVENTIONS:
Behavioral: LapSim simulator — Group B will be required to train on the LapSim simulator until they reach predefined levels of proficiency
  Other Names: Virtual reality simulator
  Arms: B

SUMMARY:
The hypothesis of this trial is to demonstrate that training junior surgeons on a virtual reality (VR) simulator in addition to didactic teaching will improve their intraoperative performance compared to those trainees who receive the traditional teaching paradigm (i.e, operating under the guidance and instruction of a consultant general surgeon).

We anticipate that the VR trained group will make less critical intraoperative errors and will perform faster than their traditionally trained colleagues.

Other study questions include:

1. Does objective assessment of fundamental abilities (FA) such as visuo-spatial ability predict intra-operative performance?
2. Do FA predict rate of learning to reach proficiency?

DETAILED DESCRIPTION:
We plan to assess up to 30 junior surgical trainees from training hospitals nationwide. All will have baseline assessment of fundamental abilities (FA) such as psychomotor, visuospatial and perceptual abilities. The trainees will then be randomised to one of two groups:

Group A-will receive the 'traditional' training programme; i.e. will receive whatever clinical training on a patient their supervising consultant deems appropriate. This is the way junior surgeons are currently trained. They will also receive the standard didactic teaching on the School for Surgeons e-learning resource.

Group B-will be assigned to the 'proficiency-based progression' training programme. These trainees will be required to train on the virtual reality (VR) simulator (Lap Sim™) for a laparoscopic cholecystectomy (LC). Trainees will have objectively set goals to reach on the simulator and will have to demonstrate proficiency before they are permitted to progress to the next, more challenging level. These supervised sessions will last no longer than one hour at a time. The proficiency measures will be predetermined errors, economy of instrument movement and economy and safety of diathermy usage.

The benchmark or 'gold standard' of proficiency will be established from the objectively assessed performance of expert consultant surgeons.

Group B will also receive the standard School for Surgeons instruction but, unlike Group A, they will have to demonstrate proficiency on the didactic module before they progress to the operating theatre.

Trainees in both the VR and traditional group will then each perform five video-recorded laparoscopic cholecystectomies at their respective training hospitals. The first three will be carried out early in the trainees rotation and the last two towards the end of the rotation. Each trainee will be supervised by a consultant surgeon for all procedures; the consultant will be ready to take over the procedure should the trainee run into difficulties.

The video recordings will be forwarded to the National Surgical Training Centre and will be assessed by two consultant surgeons blinded to the training status of the trainee.

The LC will be divided into 3 distinct phases, exposure of the cystic duct and artery plus clip placement on these structures, tissue division and finally diathermy excision of the gallbladder from the liver-bed. The different phases of the procedure will be marked, using a scoring system which will enable the observers to record whether the event or a pre-described error had or had not occurred. Senior surgeon takeover events will also be scored as errors.

ELIGIBILITY:
Inclusion Criteria:

* Consultant general surgeons who have performed > 100 laparoscopic cholecystectomies.
* General Surgical Trainees either (a) < Year 3 Higher Surgical Training (HST) , (b) < Year 3 Irish Surgical Residency Programme (ISRP) or (c) in a 'stand alone' registrar position awaiting entry to HST or ISRP.

Exclusion Criteria:

* Trainees > Year 3 HST or ISRP

Ages: 27 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
All predefined intraoperative errors committed by Group A and B while performing a supervised laparoscopic cholecystectomy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Professor Anthony Gallagher, PhD, Principal Investigator — National Surgical Training Centre, Royal College of Surgeons in Ireland
Locations (14):
- Ireland (14):
  - Portiuncula Hospital, Ballinasloe, Galway
  - Cavan General Hospital, Cavan
  - South Tipperary General Hospital, Clonmel
  - Cork University Hospital, Cork
  - South Infirmary Victoria University Hospital, Cork
  - Beaumont Hospital, Dublin
  - James Connolly Memorial Hospital, Blanchardstown, Dublin
  - St Columcilles Hospital, Loughlinstown, Dublin
  - St James Hospital, Dublin
  - University College Hospital, Galway
  - St Lukes Hospital, Kilkenny
  - Midland Regional Hospital, Portlaoise
  - Waterford General Hospital, Waterford
  - Wexford General Hospital, Wexford

REFERENCES:
- [Result] Seymour NE, Gallagher AG, Roman SA, O'Brien MK, Bansal VK, Andersen DK, Satava RM. Virtual reality training improves operating room performance: results of a randomized, double-blinded study. Ann Surg. 2002 Oct;236(4):458-63; discussion 463-4. doi: 10.1097/00000658-200210000-00008. PMID 12368674
- [Result] Gallagher AG, Lederman AB, McGlade K, Satava RM, Smith CD. Discriminative validity of the Minimally Invasive Surgical Trainer in Virtual Reality (MIST-VR) using criteria levels based on expert performance. Surg Endosc. 2004 Apr;18(4):660-5. doi: 10.1007/s00464-003-8176-z. Epub 2004 Mar 19. PMID 15026925
- [Result] Ahlberg G, Enochsson L, Gallagher AG, Hedman L, Hogman C, McClusky DA 3rd, Ramel S, Smith CD, Arvidsson D. Proficiency-based virtual reality training significantly reduces the error rate for residents during their first 10 laparoscopic cholecystectomies. Am J Surg. 2007 Jun;193(6):797-804. doi: 10.1016/j.amjsurg.2006.06.050. PMID 17512301